CLINICAL TRIAL: NCT04731116
Title: Cannabidiol Treatment for Severe and Critical COVID-19 Pulmonary Infection
Brief Title: Cannabidiol Treatment for Severe and Critical Coronavirus (COVID-19) Pulmonary Infection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, moshe yeshurun, Head BMT Unit, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0245-20-RMC
Record Dates: First submitted 2021-01-28; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CANNABIDIOL (Experimental): CANNABIDIOL 5% 3 ml twice daily for 14 days.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Oral Cannabidiol 150 mg twice daily during 14 days

SUMMARY:
Current management of COVID-19 (coronavirus) is mainly supportive, and respiratory failure from acute respiratory distress syndrome (ARDS) is the leading cause of mortality. Cytokines and chemokines are thought to play an important role in immunity and immunopathology during virus infections. Patients with severe COVID-19 have higher serum levels of pro-inflammatory cytokines (TNF-α, IL-1 and IL-6) and chemokines (IL-8) compared to individuals with mild disease or healthy controls, similar to patients with severe acute respiratory syndrome (SARS).

Cannabidiol (CBD), a nonpsychotropic ingredient of Cannabis sativa, possesses potent anti-inflammatory and immunosuppressive properties. These effects are mediated by T cell attrition and by inhibition of pro-inflammatory cytokine release (tumor necrosis factor-a, Interferon gamma, IL-1b, IL-6, and IL-17) and stimulation of anti-inflammatory cytokine production (IL-4, IL-5, IL-10, and IL-13). In a number of phase 2 trials involving more than 100 patients, our group was able to show the safety and efficacy of CBD in the prevention and treatment of graft-versus-host disease.

Based on these data, we will test the cytokine profile, safety and efficacy of CBD treatment in patients with severe and critical COVID-19 infection.

DETAILED DESCRIPTION:
Study objectives:

1. Describe the impact of CBD on the cytokine profile in patients with severe and critical COVID-19 infection.
2. Explore the safety and efficacy of CBD treatment in patients with severe and critical COVID-19 pulmonary Infection.

Methods:

This is a single center, prospective open label phase 1/2-study which will be conducted in a Corona isolation ward.

Investigational therapy:

Cannabidiol 5% dissolved in olive oil, will be given orally or through a nasogastric tube at a dose of 150 mg twice daily during 14 days or until discharge (the earliest). This dose is based on safety data generated from more than 100 transplanted patients. Treatment duration may be extended up to 28 days according to the physician discretion. In case of intolerance to the dose of 150 mg twice daily, the dose of CBD will be reduced to the maximal tolerated dose.

In the case of grade 4 side effects related to CBD or in the case of inability to provide the CBD during more the 3 days, the patient will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed novel COVID-19 infection as determined by polymerase chain reaction, or other commercial or public health assay in oropharyngeal specimen within 72 hours prior to hospitalization.
* Patients with severe disease defined as individuals with pneumonia and one or more of the following criteria:

  1. Respiratory rate ≥ 30/min.
  2. Oxygen saturation at room air less than 93%.
* Patients with critical disease defined as individuals with respiratory failure requiring mechanical ventilation
* Age18 years and older
* Informed consent has to be obtained from all patients. The patient will sign the Informed Consent Form before entering the study.
* Some patients are expected to be unable to legally consent due to critical illness, and sedation. In case a legal guardian exists, approach for consent will be made.

Exclusion Criteria:

* Allergy to CBD
* Documented infection
* Pregnant and lactating women
* Predicted clinically that there is no hope of survival
* GI intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Serum C-reactive protein (CRP) level | Daily measurement during 14 days
  Units of measurement mg%
Serum ferritin level | Daily measurement during 14 days
  Units of measurement mg%
Serum Interferon gamma-induced protein 10 (IP10) level | Daily measurement during 14 days
  Units of measurement pg/ml
Serum IL-6 level | Daily measurement during 14 days
  Units of measurement pg/ml
Serum TNF-related apoptosis-inducing ligand (TRAIL) | Daily measurement during 14 days
  Units of measurement pg/ml

SECONDARY OUTCOMES:
Study drug related adverse events | 14 days
  Number of participants with grade 3-4 study drug-related side effects as assessed by Common Terminology Criteria for Adverse Event (CTCAE) version 5.0 during treatment.
Patient adherence to the study protocol | 14 days
  Number of cannabidiol doses actually taken by the patient divided by 28 (number of planned doses)
Ratio of arterial oxygen partial pressure (PaO2) to fractional inspired oxygen (FiO2) ratio (PaO2/FiO2 ratio) for ventilated patients | 14 days
  Daily measurement of ratio of arterial oxygen partial pressure (PaO2) to fractional inspired oxygen (FiO2) ratio (PaO2/FiO2 ratio) for ventilated patients
Length of ventilation for ventilated patients | 28 days
  Number of days patient in need of mechanical ventilation
Length of stay in the ICU | 28 days
  Number of days the patient stays in ICU
Survival by day 28 | 28 days
  Patient alive (yes/no) on day 28
Remission of respiratory symptoms | 28 days
  Patient without dyspnea and saturation above 93% at room air.
Documented infections up to discharge | 28 days
  Any documented infection in addition to COVID
Sequential organ failure assistance (SOFA) score | 28 days
  Sequential organ failure assistance score calculation:range 0 to 24. A higher score is associated with higher risk of ICU mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Kagan, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeshurun M, Shpilberg O, Herscovici C, Shargian L, Dreyer J, Peck A, Israeli M, Levy-Assaraf M, Gruenewald T, Mechoulam R, Raanani P, Ram R. Cannabidiol for the Prevention of Graft-versus-Host-Disease after Allogeneic Hematopoietic Cell Transplantation: Results of a Phase II Study. Biol Blood Marrow Transplant. 2015 Oct;21(10):1770-5. doi: 10.1016/j.bbmt.2015.05.018. Epub 2015 May 30. PMID 26033282